CLINICAL TRIAL: NCT02141997
Title: A Phase 2 Study to Investigate the Safety and Efficacy of ABT-122 Given With Methotrexate in Subjects With Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate
Brief Title: A Study to Investigate the Safety and Efficacy of ABT-122 Given With Methotrexate in Subjects With Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-963; 2013-004019-37 (EudraCT Number)
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
Keywords: efficacy; Methotrexate; safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; ABT-122

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Adalimumab 40 mg EOW (Active Comparator): Adalimumab 40 mg every other week (EOW) for 11 weeks.
  Interventions: Biological: adalimumab
- ABT-122 60 mg EOW (Experimental): ABT-122 60 mg every other week (EOW) for 11 weeks.
  Interventions: Biological: ABT-122
- ABT-122 120 mg EOW (Experimental): ABT-122 120 mg every other week (EOW) for 11 weeks.
  Interventions: Biological: ABT-122
- ABT-122 120 mg EW (Experimental): ABT-122 120 mg every week (EW) for 11 weeks.
  Interventions: Biological: ABT-122

INTERVENTIONS:
Biological: adalimumab — adalimumab administered as subcutaneous injection every other week (EOW)
  Other Names: Humira
  Arms: Adalimumab 40 mg EOW
Biological: ABT-122 — ABT-122 administered as subcutaneous injection every other week (EOW)
  Arms: ABT-122 120 mg EOW; ABT-122 120 mg EW; ABT-122 60 mg EOW

SUMMARY:
This study is a Phase 2 randomized, double-blind, double-dummy, parallel-group study designed to assess the safety, tolerability, efficacy, pharmacokinetics and immunogenicity of multiple doses of ABT 122 in subjects with active rheumatoid arthritis (RA) who are inadequately responding to methotrexate (MTX) treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, 18 years of age or older.
2. Diagnosis of RA based on the 2010 American College of Rheumatology (ACR)/European League against Rheumatism (EULAR) criteria (as defined in the definition of terms).
3. Rheumatoid Arthritis (RA) diagnosis at least 3 months from the date of first Screening.
4. Have active RA defined by minimum disease activity criteria:

   * ≥ 6 Swollen joints (based on 66 joint counts) at screening and baseline visits.
   * ≥ 6 Tender joints (based on 68 joint counts) at screening and baseline visits.
   * hsCRP> ULN OR positive for both Rheumatoid Factor (RF) and Anti-Cyclic Citrullinated Peptide (Anti-CCP) Antibody levels at screening.
5. Inadequate response to Methotrexate (MTX) treatment defined as oral or parenteral treatment ≥ 3 months with an unchanged mode of application and stable prescribed MTX dose for at least 4 weeks prior to baseline of ≥ 10mg/week and < the upper limit of the applicable approved local label. Subject can also be on stable doses of sulfasalazine and/or hydroxychloroquine, so long as they are also on methotrexate.

Exclusion Criteria:

1. Subject has previous exposure to Humira, other Tumor necrosis factor (TNF) inhibitors or other biological DMARDs.
2. Current treatment with traditional oral Disease modifying antirheumatic drugs (DMARDs) (except for concomitant treatment with sulfasalazine and/or hydroxychloroquine in addition to MTX). Oral DMARDs must be washed out 5 times the mean terminal elimination half-life of a drug apart from MTX prior to Day 1.

   • Subject could have been exposed to prior Janus kinase (JAK) inhibitors so long as they have been off therapy for 5 half-lives.
3. Stable prescribed dose of oral prednisone or prednisone equivalent > 10 mg/day within the 30 days of first dose of study drug.
4. Intra-articular or parenteral administration of corticosteroids in the preceding 4 weeks of first dose of study drug. Inhaled corticosteroids for stable medical conditions are allowed.
5. Laboratory values of the following at the Screening Visit:

   * Confirmed hemoglobin < 9 g/dL for males and < 8.5 g/dL for females,
   * Absolute neutrophil count (ANC) < 1500 mm^3,
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 × the upper limit of normal (ULN) or bilirubin ≥ 3 mg/dL,
   * Serum creatinine > 1.5 × the ULN,
   * Platelets < 100,000 cells/[mm3] (10^9/L),
   * Clinically significant abnormal screening laboratory results as evaluated by the Investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Mansikka, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Genovese MC, Weinblatt ME, Aelion JA, Mansikka HT, Peloso PM, Chen K, Li Y, Othman AA, Khatri A, Khan NS, Padley RJ. ABT-122, a Bispecific Dual Variable Domain Immunoglobulin Targeting Tumor Necrosis Factor and Interleukin-17A, in Patients With Rheumatoid Arthritis With an Inadequate Response to Methotrexate: A Randomized, Double-Blind Study. Arthritis Rheumatol. 2018 Nov;70(11):1710-1720. doi: 10.1002/art.40580. Epub 2018 Oct 10. PMID 29855172
- See also: Humira Prescribing info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 30-day screening period.
Period: Overall Study
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Started | 56 | 55 | 56 | 55
Completed | 53 | 49 | 53 | 54
Not Completed | 3 | 6 | 3 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Participant noncompliance | 1 | 0 | 0 | 0
Not completed — Withdrew consent | 1 | 0 | 3 | 0
Not completed — Other | 1 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW | Total
Number analyzed (Participants) | 56 | 55 | 56 | 55 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.36) | 55.2 (11.81) | 53.5 (13.00) | 55.6 (12.34) | 55.5 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 49 | 45 | 181
  Male | 14 | 10 | 7 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Response defined as at least 20% reduction (improvement) compared with baseline in tender joint count (TJC68), swollen joint count (SJC66), and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, patient's global assessment of disease activity (PtGA); physician's global assessment of disease activity (PGA), Health Assessment Questionnaire - Disability Index (HAQ-DI), and high-sensitivity C-reactive protein (hsCRP). Last observation carried forward (LOCF) was used for missing data (only post-baseline values were carried forward).
Time Frame: Baseline (Day 1) and Week 12
Population: Full analysis set (FAS) defined as all randomized participants with at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 55
percentage of participants | 73.2 | 65.5 | 76.8 | 81.8
Statistical Analysis 1: Comparison: Adalimumab 40 mg EOW vs ABT-122 60 mg EOW; P-value calculated using 1-sided Fisher's Exact test; Test type: Superiority or Other; p = 0.863, Fisher Exact
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EOW; P-value calculated using 1-sided Fisher's Exact test; Test type: Superiority or Other; p = 0.414, Fisher Exact
Statistical Analysis 3: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; P-value calculated using 1-sided Fisher's Exact test; Test type: Superiority or Other; p = 0.196, Fisher Exact

2. Secondary Outcome: Change in Disease Activity Score 28 With High Sensitivity C-Reactive Protein (DAS28 [hsCRP])
Description: The DAS28 (hsCRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hsCRP, and general health are included in the DAS28 (hsCRP) score. Scores range from 0 to 10: a score >5.1 indicates high disease activity, a score <3.2 indicates low disease activity, and a score <2.6 indicates clinical remission. A negative change from baseline represents improvement. n=the number of participants with evaluable data at each time point. LOCF was used (only post-baseline values were carried forward).
Time Frame: Baseline, Weeks 2, 4, 6, 8, and 12
Population: Subjects in the FAS with a baseline value and at least 1 post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 55
units on a scale
  Week 2 (n=54,53,55,53) | -1.43 [-1.71 to -1.15] | -1.26 [-1.54 to -0.97] | -1.80 [-2.08 to -1.52] | -1.69 [-1.97 to -1.41]
  Week 4 (n=56,55,56,55) | -1.86 [-2.17 to -1.55] | -1.66 [-1.97 to -1.34] | -2.08 [-2.39 to -1.78] | -2.15 [-2.46 to -1.84]
  Week 6 (n=56,55,56,55) | -2.28 [-2.60 to -1.96] | -1.83 [-2.16 to -1.51] | -2.39 [-2.71 to -2.07] | -2.41 [-2.74 to -2.09]
  Week 8 (n=56,55,56,55) | -2.32 [-2.64 to -2.00] | -1.98 [-2.31 to -1.65] | -2.60 [-2.93 to -2.28] | -2.58 [-2.91 to -2.25]
  Week 12 (n=56,55,56,55) | -2.44 [-2.75 to -2.12] | -2.06 [-2.38 to -1.74] | -2.64 [-2.95 to -2.33] | -2.67 [-2.98 to -2.35]

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Response defined as at least 50% reduction (improvement) compared with baseline in tender joint count (TJC68), swollen joint count (SJC66), and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, PtGA; PGA, HAQ-DI, and hsCRP. LOCF was used (only post-baseline values were carried forward).
Time Frame: Baseline (Day 1) and Week 12
Population: Participants in the FAS population with a baseline value and at least 1 post-baseline value
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 54
percentage of participants | 51.8 | 34.5 | 48.2 | 48.1

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Response defined as at least 70% reduction (improvement) compared with baseline in tender joint count (TJC68), swollen joint count (SJC66), and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, PtGA; PGA, HAQ-DI, and hsCRP. LOCF was used (only post-baseline values were carried forward).
Time Frame: Baseline (Day 1) and Week 12
Population: Participants in the FAS population with a baseline value and at least 1 post-baseline value
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 55
percentage of participants | 23.2 | 23.6 | 19.6 | 36.4

5. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) or Clinical Remission (CR) Based on DAS28 (hsCRP) at Week 12
Description: The DAS28 (hsCRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hsCRP, and general health are included in the DAS28 (hsCRP) score. Scores range from 0 to 10: a score >5.1 indicates high disease activity, a score <3.2 indicates low disease activity, and a score <2.6 indicates clinical remission. LDA is defined as a DAS28 (hsCRP) score from 2.6 to < 3.2 at Week 12. CR is defined as a DAS28 (hsCRP) score < 2.6 at Week 12. LOCF was used (only post-baseline values were carried forward).
Time Frame: Week 12
Population: Participants in the FAS population with a baseline value and at least 1 post-baseline value
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 55
percentage of participants | 50.0 | 34.5 | 53.6 | 54.5

6. Secondary Outcome: Percentage of Participants Achieving CR Based on DAS28 (hsCRP) at Week 12
Description: The DAS28 (hsCRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hsCRP, and general health are included in the DAS28 (hsCRP) score. Scores range from 0 to 10: a score >5.1 indicates high disease activity, a score <3.2 indicates low disease activity, and a score <2.6 indicates clinical remission. CR is defined as a DAS28 (hsCRP) score < 2.6 at Week 12. LOCF was used (only post-baseline values were carried forward).
Time Frame: Week 12
Population: Participants in the FAS population with a baseline value and at least 1 post-baseline value
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 55
percentage of participants | 32.1 | 23.6 | 39.3 | 41.8

7. Secondary Outcome: Percentage of Participants Achieving LDA or CR Based on Clinical Disease Activity Index (CDAI) at Week 12
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. LDA is defined as a CDAI score from 2.8 to ≤ 10 at Week 12. CR is defined as a CDAI score ≤ 2.8 at Week 12. LOCF was used (only post-baseline values were carried forward).
Time Frame: Week 12
Population: Participants in the FAS population with a baseline value and at least 1 post-baseline value
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 55
percentage of participants | 42.9 | 36.4 | 44.6 | 54.5

8. Secondary Outcome: Percentage of Participants Achieving CR Based on Clinical Disease Activity Index (CDAI) at Week 12
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. CR is defined as a CDAI score ≤ 2.8 at Week 12. LOCF was used (only post-baseline values were carried forward).
Time Frame: Week 12
Population: Participants in the FAS population with a baseline value and at least 1 post-baseline value
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Number analyzed (Participants) | 56 | 55 | 56 | 55
percentage of participants | 8.9 | 7.3 | 10.7 | 10.9

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 21 weeks); serious adverse events (SAEs) were collected from the time informed consent was obtained (25 weeks).
Description: A TEAE is defined as any AE with onset or worsening reported by a participant from the time that the first dose of study drug is administered until 70 days have elapsed following discontinuation of study drug administration. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Adalimumab 40 mg EOW | ABT-122 60 mg EOW | ABT-122 120 mg EOW | ABT-122 120 mg EW
Serious Adverse Events (participants affected / at risk) | 0/56 | 2/55 | 0/56 | 2/55
Other Adverse Events (participants affected / at risk) | 12/56 | 11/55 | 11/56 | 10/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg EOW (N=56) | ABT-122 60 mg EOW (N=55) | ABT-122 120 mg EOW (N=56) | ABT-122 120 mg EW (N=55)
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg EOW (N=56) | ABT-122 60 mg EOW (N=55) | ABT-122 120 mg EOW (N=56) | ABT-122 120 mg EW (N=55)
DIARRHOEA (Gastrointestinal disorders) | 2 | 3 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 2 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2 | 2
NASOPHARYNGITIS (Infections and infestations) | 3 | 2 | 1 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 4
URINARY TRACT INFECTION (Infections and infestations) | 1 | 5 | 1 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 3 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 3 | 0
HEADACHE (Nervous system disorders) | 0 | 3 | 2 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 2 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
HYPERTENSION (Vascular disorders) | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.